CLINICAL TRIAL: NCT06926985
Title: An Exploratory Clinical Study of the Safety and Efficacy of Anti-CD19/BCMA Chimeric Antigen Receptor NK Cell Injection in the Treatment of IgA Nephropathy
Brief Title: An Exploratory Clinical Study of Anti-CD19/BCMA Chimeric Antigen Receptor NK Cell Injection in the Treatment of IgA Nephropathy
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Due to limitation of production capacity
Sponsor: Jieyang People's Hospital (Other)
Responsible Party: Principal Investigator, Qinghua Liu, Professor, Jieyang People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025002
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: IgA Nephropathy (IgAN)
Keywords: IgA Nephropathy; CD19 BCMA CAR NK; SLE
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19 BCMA CAR NK cells (Experimental)
  Interventions: Biological: anti-CD19/BCMA CAR NK cells

INTERVENTIONS:
Biological: anti-CD19/BCMA CAR NK cells — Patients will receive Fludarabine and Cyclophosphamide on day -5, -4, and -3. Multiple doses of anti-CD19/ BCMA CAR NK cells will infused using the dose-escalation strategy.

SUMMARY:
A single arm, open-label pilot study is designed to evaluate the safety and effectiveness of anti-CD19/BCMA CAR NK cells (KN5601) in patients with IgA nephropathy

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old and ≤ 70 years old, male or female;
2. IgA nephropathy confirmed by pathological biopsy of renal biopsy;
3. All females of childbearing potential must use effective contraception during treatment and for 90 days after the last dose of treatment. In addition, subjects must not donate eggs during the study and for at least 90 days after the last dose of treatment;
4. Urine total protein/urine creatinine ratio (UPCR) ≥ 500 mg/g and estimated glomerular filtration rate (eGFR) > 20 ml/min/1.73m2 during the screening period

Exclusion Criteria:

1. Subjects with IgA nephropathy with rapidly progressive renal function, pathological manifestations include extensive crescent formation and necrotic vascular lesions in the glomeruli;
2. Secondary IgA nephropathy;
3. Subjects do not take medication regularly or stop taking medication during treatment;
4. Individuals with known severe allergic reactions, hypersensitivity, contraindication to any medications during the trial (cyclophosphamide, fludarabine, tozumabs), or subjects with a history of severe allergic reactions;
5. Subjects with active infection (except simple urinary tract infection and bacterial pharyngitis), or currently receiving intravenous antibiotic treatment, or subjects who have received intravenous antibiotic treatment within 1 week before KN5601 infusion;
6. Subjects with acquired and congenital immunodeficiency diseases;
7. Subjects with grade III or IV heart failure (NYHA classification);
8. History of epilepsy or other central nervous system (CNS) diseases;
9. History of severe herpes infection, such as herpes encephalitis, ocular herpes, or disseminated herpes; signs of herpes or varicella-zoster virus infection (especially chickenpox, herpes zoster) within 12 weeks prior to screening;
10. History of other primary malignant tumors except:
11. Cured non-melanoma skin cancer by surgical excision, for example basal cell carcinoma (BCC) ;
12. Cured primary malignant tumors, such as cervical cancer, superficial bladder cancer, breast cancer
13. Has a history of any clinically significant cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urinary, pulmonary, neurological, dermatologic, psychiatric, and renal disease or other significant disease that precludes KN5601 administration (as determined by the investigator), except IgA nephropathy;
14. Females who are pregnant, lactating, or planning a pregnancy within six months;
15. Subjects who have received other clinical trial treatment within 3 months;
16. Subjects who have received B cell-targeted drug therapy within 1 months before enrollment;
17. Any abnormal laboratory test results judged by the investigator to be clinically significant and prevent the subject from participating in the study. Laboratory test values that are out of range and not of clinical significance will not be considered as exclusion criteria;
18. Any situation judged by the investigators that may increase the risk of the subjects or interfere with the clinical trial outcome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicity (DLT) | up to 52 weeks after infusion
  To characterize the safety of CD19 CAR NK Cells (KN5601) for IgA Nephropathy
Incidence of Treatment Emergent Adverse Events (TEAEs) | up to 52 weeks after infusion
  To characterize the safety of CD19 CAR NK Cells (KN5601) for IgA Nephropathy

SECONDARY OUTCOMES:
The complete response rate | 52 weeks after infusion
  To characterize the efficacy of CD19 CAR NK Cell (KN5601) for for IgA Nephropathy
The partial response rate | 48 weeks after infusion
  To characterize the efficacy of CD19 CAR NK Cell (KN5601) for for IgA Nephropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Jieyang People's Hospital, Jieyang, Guangdong, China